CLINICAL TRIAL: NCT04814264
Title: Pilot Study of Sex-matched vs. Sex-mismatched Red Blood Cell Transfusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michelle Zeller, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sex_MATTERS
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Blood Transfusion
Keywords: Blood; Transfusion; Intensive care; Sex-matched; Sex-mismatched
MeSH Terms: interventions — Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: Multicentre, pilot randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blood bank staff will be blinded to the treatment allocation schedule and the use of random block sizes in the allocation schedule will ensure that they are not aware of which treatment will be assigned next. The clinical staff will be blinded to the intervention. The study biostatistician will be blinded to treatment allocation for any analyses performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sex-matched red blood cell transfusion (Experimental): All patients will receive red blood cells (RBCs) that are ABO and Rh compatible as per routine blood bank practices. In addition to routine compatibility, subjects in this arm will receive blood that is matched to their sex (donor and recipient sex are the same). Patients in this arm will receive RBCs matched to their sex until discharge from hospital or death.
  Interventions: Biological: Red blood cells
- Sex-mismatched red blood cell transfusion (Experimental): All patients will receive red blood cells (RBCs) that are ABO and Rh compatible as per routine blood bank practices. In addition to routine compatibility, subjects in this arm will receive blood that is not matched to their sex (donor and recipient sex are not the same). Patients in this arm will receive RBCs mismatched to their sex until discharge from hospital or death.
  Interventions: Biological: Red blood cells

INTERVENTIONS:
Biological: Red blood cells — All transfused red blood cells will be obtained from Canadian Blood Services and will be the standard red blood cell products currently provided in Canada.

SUMMARY:
Blood transfusion is common for patients in hospital, especially for those in intensive care. Patients receive blood that is matched to them based on their blood group (A, B, AB, O), but not based on sex. This means male or female patients may receive male or female blood. There is some evidence to suggest that giving male patients female blood and female patients male blood (sex-mismatched blood) may be harmful. The investigators think giving males only male blood and females only female blood (sex-matched blood) will be better for the patients and improve their survival. To test this, the study team will randomly give 50% of intensive care patients who require blood only sex-mismatched blood and 50% of intensive care patients only sex-matched blood for their entire hospital stay. Then, health data of patients will be collected to see if either group does better after transfusion. Before this is done as a large study with thousands of patients, it will be attempted as a smaller pilot study with a few hundred patients to be sure the processes suggested make sense and are possible for hospitals and for the blood supplier to follow.

DETAILED DESCRIPTION:
Blood transfusion is one of the most common procedures performed during hospitalization. Approximately 85 million red blood cell (RBC) units are transfused globally each year. RBC units are matched for blood groups but matching for other donor characteristics such as sex, is not considered. By the current standard of care, female or male patients can receive RBCs from male or female donors. However, accumulating data suggests that sex-mismatched transfusions may be harmful.

Sex-mismatched transfusions and transplantations have been associated with poor outcomes. Plasma from female donors is associated with an increased risk of transfusion related acute lung injury (TRALI); sex-mismatched heart transplantation is associated with increased transplant-associated mortality; and stem cell transplants from female donors are associated with worse outcomes.

Anemia is common during critical illness and 20-40% of critically ill patients require a mean of two to five RBC units during admission to the intensive care unit (ICU). Once a patient receives more than six RBC units, virtually all patients (>97%) will have received at least one sex-mismatched RBC. The population of transfused ICU adult patients is already at high risk of death, with a demonstrated 90-day all-cause mortality of 35-37% based on the ABLE study, and in-hospital mortality of 24-34% (institutional data). Thus, new supportive care strategies are needed to improve outcomes of this highly vulnerable patient group.

Transfusion data linked to donor sex spanning a 6-year period was previously analyzed. Using a careful analysis that controlled for covariates and stratified on time-dependent and fixed variables, 25,219 transfusion recipients were retrospectively analyzed and a significant association between male to female RBC transfusions and death [hazard ratio (HR) 1.31, 95% confidence interval (CI) 1.02-1.69] was found. A trend towards higher mortality was also noted with female to male RBCs (HR 1.13: 95% CI 0.92-1.39), and with sex-mismatched vs. sex-matched RBCs overall (HR 1.23: 95% CI 1.04-1.45). These findings suggest that matching RBC transfusions for sex can reduce mortality in ICU patients.

The investigators hypothesize that donor-recipient sex-matched RBC transfusions are associated with improved survival in hospital compared to sex-mismatched RBC transfusions. Sex-matched RBC transfusions may represent an important, readily implementable advance in supportive care of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18)
* Admitted to the intensive care unit
* Requiring a red blood cell transfusion

Exclusion Criteria:

* Requiring a specific red blood cell unit or unit not readily available (e.g., phenotypically matched, rare blood, washed, complex red blood cell antibodies, etc.)
* Massively bleeding (i.e. ≥4 units of blood ordered, or Massive Hemorrhage Protocol initiated, or an urgent blood request made)
* Biological sex unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome - Missing randomization rate (%) | From date of study initiation at each site until date the final patient is randomized, approximately 8 months.
  Feasibility of randomizing consecutive eligible patients in the intensive care unit who require blood transfusion. Data collected electronically at monthly intervals. Missing randomization rate calculated by taking the number of eligible patients not randomized divided by the total number of eligible patients × 100%.
Feasibility outcome - Recruitment compliance (%) | From date the first patient is randomized until 30 days after the final patient is randomized.
  Number of recruitments that are compliant out of all randomizations. Reasons for recruitment non-compliance include: (a) duplicate randomization; (b) entering incorrect identification number into the randomization program; (c) patient randomized not admitted to ICU; and, (d) randomized ICU patients not transfused. Data collected electronically at monthly intervals. Frequency of recruitment compliance calculated by taking the number of recruitments that are compliant divided by the total number of patients randomized ×100%.
Feasibility outcome - Protocol adherence (%) | From date the first patient is randomized until 30 days after the final patient is randomized.
  The proportion of patients in the intervention arms who receive all red blood cell transfusions as sex-matched/sex-mismatched out of all transfused per intervention arm. Data collected electronically at monthly intervals. Percentage protocol adherence rate calculated by taking the number of patients in the intervention arm who receive all RBC transfusions as sex-matched or mismatched divided by the total number of transfused patients in the intervention arm x 100%.

OTHER OUTCOMES:
Data collection outcome - Ability to provide timely monthly reports | From date of study initiation at each site until 30 days after the final patient is randomized.
  Ability of each participating site to provide timely monthly reports to monitor inventory levels and mortality outcomes.
Data collection outcome - Rate of post-randomization exclusions (%) | From date the first patient is randomized until 30 days after the final patient is randomized.
  Rate of post-randomization exclusions calculated by taking the number of patient exclusions post randomization divided by the total number randomized x 100%.
Patient important clinical outcomes - In-hospital mortality (%) | From date the first patient is randomized until 30 days after the final patient is randomized.
  In-hospital mortality calculated by taking the number of deaths in hospital divided by the total number randomized x 100%.
Patient important clinical outcomes - Time to death (days) | From date of patient randomization until the date of death from any cause while in hospital, assessed up to 30 days after the final patient is randomized.
  Time to death in days, only applicable to patients who die while in hospital.
Patient important clinical outcomes - Hemoglobin increment (g/L) | From date of patient randomization until the date of discharge from hospital or date of death from any cause, whichever comes first, assessed up to 30 days after the final patient is randomized.
  Hemoglobin increment calculated by taking the post-transfusion hemoglobin value minus the pre-transfusion hemoglobin value.
Patient important clinical outcomes - Creatinine level and increment (umol/L) | From date of patient randomization until the date of discharge from hospital or date of death from any cause, whichever comes first, assessed up to 30 days after the final patient is randomized.
  Creatinine increment calculated by taking the post-transfusion creatinine value minus the pre-transfusion creatinine value.
Patient important clinical outcomes - ICU/hospital length of stay (days) | From date of patient randomization until the date of discharge from hospital or date of death from any cause, whichever comes first, assessed up to 30 days after the final patient is randomized.
  Days admitted to ICU and/or hospital.
Patient important clinical outcomes - Number/type of transfused products (unit/volume) | From date of patient randomization until the date of discharge from hospital or date of death from any cause, whichever comes first, assessed up to 30 days after the final patient is randomized.
  Number of units and/or volume and type of blood products/plasma derivatives transfused.
Patient important clinical outcomes - Number/type of transfusion reactions | From date of patient randomization until the date of discharge from hospital or date of death from any cause, whichever comes first, assessed up to 30 days after the final patient is randomized.
  Number and type of transfusion reactions reported.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Zeller, MD, Principal Investigator — McMaster University
Locations (5):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066